# FRIDs and fall risk among older adults - protocol

# Title:

Potential Fall-Risk-Increasing Drugs and falls in community-dwelling older adults: A prospective cohort study

# Registration

Clinicaltrials.gov Identifier: NCT05169476

# Document date

12-23-2021

**Funding** 

This research will be funded by The Department of Geriatrics, Aalborg University Hospital, Den-

mark, The Department of Clinical Medicine, Aalborg University, Denmark, The municipality of

Hjørring, Denmark and by external funding. The external funding sources will have no role in the

design of this study, during its execution, analyses, interpretation of data or decision to submit re-

sults.

**Authors** 

Corresponding author:

Silas Zacharias Clemmensen, MS

Department of Geriatrics, Aalborg University Hospital, Denmark

Department of Health Science and Technology, Aalborg University, Aalborg, Denmark

E-mail: silas.clemmensen@rn.dk

Jens Eg Nørgaard, MSc

Department of Geriatrics, Aalborg University Hospital, Denmark

Department of Clinical Medicine, Aalborg University, Aalborg, Denmark

E-mail: jens.noergaard@rn.dk

Gustav Valentin Gade, MD, PhD

Department of Geriatrics, Aalborg University Hospital, Denmark

Department of Clinical Medicine, Aalborg University, Denmark.

E-mail: gustav.soerensen@rn.dk

Martin Grønbech Jørgensen, MSc, PhD, Assistant Professor

Department of Geriatrics, Aalborg University Hospital, Denmark.

E-mail: mgj@rn.dk

2

Nadja Albertsen, MD

Department of Geriatric Medicine, Aalborg University Hospital, Aalborg, Denmark Arctic Health Research Centre, Aalborg University Hospital, Aalborg, Denmark Department of Clinical Medicine, Aalborg University, Aalborg, Denmark <a href="mailto:n.albertsen@rn.dk">n.albertsen@rn.dk</a>

Stig Andersen, MD, PhD, Professor.

Department of Geriatrics, Aalborg University Hospital, Denmark and Arctic Health Research Centre, Aalborg University Hospital, Aalborg, Denmark Department of Clinical Medicine, Aalborg University, Denmark.

E-mail: <u>lasa@rn.dk</u>

# **Sponsor contact information**

#### Study sponsor:

Department of Geriatrics, Aalborg University Hospital, Denmark.

#### Contact name:

Stig Andersen, MD, PhD, Professor. E-mail: lasa@rn.dk

#### Address:

Geriatrisk afdeling, Gl. Rød bygn. 6, 2. Etage

Aalborg Universitetshospital, Syd, Hobrovej 18-22, 9000 Aalborg

#### Introduction

Falls in community-dwelling older adults are a major public health issue with an annual incidence of approximately 30% among adults aged  $\geq$ 65 years increasing to 32-42% among those aged  $\geq$ 75 years (1). In addition, the number of fallers is expected to increase in the future since the proportion of older people over 60 years is increasing worldwide (2). In Europe, the most frequent reason for older adults to contact an emergency department is due to falls - accounting for 50% of the total contacts (3). Even though most of the falls result in minor injuries, an increasing proportion leads to fractures or hospitalization. Furthermore, consequences of falls include increased morbidity and mortality along with loss of independence, which may lead to early institutionalization (1,4,5). Finally, the increasing number of fallers also leads to increased financial burden on the health care system (6).

Although some falls have a single obvious reason, most falls have a multifactorial aetiology such as previous falls, advanced age, cognitive impairment, environmental risks, hazardous activities, along with presence of chronic disease, muscle weakness, gait and balance disorders, and medication use (1,4,7–13). Recently, The European Geriatric Medicine Society (EuGMS) Task and Finish Group published a consensus paper classifying 14 medication classes as fall-risk-increasing drug (FRID) (14). Most of them were psychotropics, but several new possible FRIDs were identified. However, the group did not reach consensus on 17 medication classes as potential FRIDs (antihypertensives, cardiac glycosides, antiarrhythmics, gastrointestinal agents, central nervous system agents, chemotherapeutics, hypoglycaemics, fluoroquinolones, corticosteroids, and nonsteroidal anti-inflammatory drugs). This was substantiated by the studies presented for the panellists being heterogenous due to various settings, different cohorts of older adults as well as unclear descriptions of the medication and falls ascertainment methods. Hence, the evidence was insufficient to attain consensus.

This is consistent with the current gap in the literature with only a few studies investigating fall risk related to these types of drugs (15–17). Moreover, the group advocated for a higher research quality in primary studies due to issues with precise definitions of target medications and falls as well as lack of controlling for confounders (14,18). Therefore, to achieve a better understanding of these 17 medication classes as potential FRIDs, more studies taking these issues into account are warranted.

#### Primary objective:

To examine the association between use of the potential FRIDs and falls rate with a 1-year followup in a cohort of community-dwelling older adults, aged 75 years or more.

#### **Study methods**

#### Study design and sample size:

This prospective cohort study builds on previous data from the PREFALL study conducted in cooperation with Hjørring Municipality, Denmark (19). A pre-registered protocol on the PREFALL study was accepted at Clinicaltrials.gov (NCT03608709) on 01/08/2018 (20). The study recruited participants from 14/06/2018 to 18/07/2019 and had a 1-year follow-up period. The sample size was derived without a recommended power calculation; hence, the sample size builds on feasible recruitment within the 13 months inclusion period granted by the municipality due to economical and administrative reasons.

#### Timing of final analysis:

All study data were accessible from the PREFALL study before the completion of this protocol. Therefore, a detailed statistical analysis plan for this study was prepared before any outcome analysis was conducted to provide transparency on the intended and pre-planned analysis. This is prespecified later in the protocol.

#### Study population and setting

The participants were community-dwelling aged 75 or more. Participants were excluded if they had 1) a dementia diagnosis; 2) acute illness defined by the presence of a participant-reported experience of illness within 7 days before inclusion affecting their ability to participate in social activities outside their homes; 3) inability to understand Danish; 4) Unable to stand unassisted for one minute. Support was defined by any assistive devices or help from another person. In Denmark, municipalities develop and initiate prophylactic and health-promoting initiatives for senior citizens (22). Thus, the participants were recruited through preventive home visits (PHV), senior activity centres (SAC), along with senior clubs and associations in Hjørring Municipality, Northern Jutland, Denmark. For PHVs, all the community-dwellers aged 75+ years who accepted the invitation to PHV were assessed for eligibility and included consecutively. For SACs, senior clubs, and senior associations, participants were conveniently recruited by oral study presentations since a

consecutive sampling method was not possible due to varying attendees each day. Lastly, recruitment videos were transmitted by the local televisions channel along with ads in newspapers and social media. For a more detailed description of the study setting and recruitment, the investigators refer to the PREFALL study (19).

#### Follow-up:

Follow-up time will be defined as the time from inclusion until death, withdrawal, or end of the study at the 18/07/2020. A summary of the participants' loss to follow-up will be presented with reasons and baseline characteristics to describe the adequacy of follow-up.

#### Baseline characteristics:

Data collection was performed at baseline and based on a multifactorial falls risk test battery including various physical tests (static balance under dual-task conditions, grip- and lower limb strength, reaction time of lower limbs and gait speed); self-report questionnaire on sociodemographic characteristics, frailty, nutrition, disability, fear of falling, health-related quality of life, depressive symptoms, several physical symptoms, cognitive tests; and reporting of comorbidities (23). The participants' comorbidities were obtained from the participants' hospital records and the diagnoses were indexed according to the International Classification of Diseases 10<sup>th</sup> revision (ICD-10). For a more detailed description of physical test and self-report questionnaire and their rationale, the investigators refer to the PREFALL study (19).

#### Baseline medication:

To determine the participants' medications at inclusion, the investigators consulted the national Shared Medication Record (SMR). The SMR is a national registry of current medication use and pharmacy records of prescriptions to each citizen in Denmark. Any physician involved in the patients' clinical course has access to the SMR data and all details of each prescription and the date of the latest medication reconciliation are provided (24). For each participant all medication registered in SMR at baseline was documented and indexed according to the WHO-recommended anatomical therapeutic chemical (ATC) medication classification system. The potential FRIDs which will be investigated in this study are: Beta-blockers (C07A); angiotensin-converting enzyme (ACE) inhibitors (C09A); calcium channel blockers (C08); cardiac glycosides (C01A); antiarrhythmic drugs (C01B); laxatives (A06A); proton pump inhibitors (A02BC); antiparkinson drugs (N04); acetylcholinesterase inhibitors (N06DA); beta blocker eye drops (S01ED); corticosteroid (H02A); oral

hypoglycaemic drugs (A10B); vitamin D (A11CC05); nonsteroidal anti-inflammatory (NSAID) drugs (M01A); fluoroquinolones (J01MA); and antineoplastic agents (L01).

#### Confounding covariates:

Many different risk factors and predictors for falls in older adults have been described previously and classified into different domains: sociodemographic, medical conditions, psychological, balance and mobility, and medication use (4,25,26). All these risk factors are possible confounders to the potential FRIDS; hence, the following a priori list specifies the confounding variables to be adjusted for in the multivariate regression model:

- Age (5,8).
- Sex (4).
- History of previous falls (19,27,28).
- The comorbidity related to the potential FRID to adjust for confounding by indication (18).
- Fear of falling using Short Falls Efficacy Scale-International 7-item (4,27–30).
- Gait speed measured with a 4-meter walk test (31–33).
- Cognitive impairment estimated by the Orientation-Memory-Concentration test performed over the telephone (4,27,33,34).
- Frailty using the Tilburg Frailty Indicator (35).
- Physical and instrumental disability in activities of daily living using the Vulnerable Elders Survey 13 (4,32,33,36).
- Depressive symptoms using Geriatric Depression Scale 4 item, a depression diagnosis or prescription of any antidepressants (4,16,27,28).
- Use of benzodiazepines, benzodiazepines derivatives or non-benzodiazepines (Z-drugs) (16,37).
- Use of opioids (15,38).

### Statistical analysis

#### Outcome:

The primary outcome is fall rate per person-year. Fall rate will be calculated as the total number of falls divided by length of follow-up in years. A fall was defined as "an unexpected event in which the participants come to rest on the ground, floor, or lower lever" (39). Falls were recorded

prospectively with daily fall calendars with a monthly reporting and validated by a phone call if a fall was registered. If the calendar was not received within 14 days after deadline, the participant was contacted to retrieve the missing data.

#### Statistical methods:

A flowchart will be given to illustrate the flow of participants through the study including number of participants with and without falls. The participants' baseline characteristics and follow-up time will be summarised using descriptive statistics. Continuous variables will be summarized using medians with interquartile range, and categorical variables will be presented using counts and percentage proportions. Furthermore, the number of participants with missing data for the outcome, baseline characteristics, and confounding covariates will be presented. Then, missing data will be handled with multiple imputation methods. Finally, a univariate and multivariate Poisson regression model will be used to specify the association (expressed as incidence rate ratio, IRR) between the potential FRID and the rate of falls. For each potential FRID, a multivariate Poisson regression model will be performed adjusting for the medical indication of each drug and all other confounders from the a priori list. However, the Poisson regression model will only be performed for the potential FRID if more than 5 participants have a prescription registered at baseline. P-values lower than 0.05 will be considered as statistically significant. All statistical analyses will be carried out using R, version 4.0.2, (R Foundation).

#### Dissemination and reporting

The investigators want to publish the study in peer-reviewed journals in English. The reporting of the study will follow the Strengthening the Reporting of Observational studies in Epidemiology (STROBE) statement.

#### **References:**

- 1. Masud T, Robert OM. Epidemiology of falls. 2001;3–7.
- 2. Organization WH. WHO Global report on Falls Prevention in Older Age. Community Health. 2007.
- 3. EuroSafe. Injuries in the European Union, Summary on Injury Statistics 2012-2014. Amsterdam; 2016.
- 4. Deandrea S, Lucenteforte E, Bravi F, Foschi R, La Vecchia C, Negri E. Risk factors for falls in community-dwelling older people: A systematic review and meta-analysis. Epidemiology. 2010 Sep;21(5):658–68.
- 5. Rubenstein LZ. Falls in older people: Epidemiology, risk factors and strategies for prevention. Age Ageing. 2006;35(SUPPL.2):37–41.
- 6. Scuffham P, Chaplin S, Legood R. Incidence and costs of unintentional falls in older people in the United Kingdom. J Epidemiol Community Health. 2003;57(9):740–4.
- 7. Ambrose AF, Paul G, Hausdorff JM. Risk factors for falls among older adults: A review of the literature. Maturitas [Internet]. 2013;75(1):51–61. Available from: http://dx.doi.org/10.1016/j.maturitas.2013.02.009
- 8. Tinetti ME, Speechley M, Ginter SF. Risk factors for falls among elderly persons living in the community. Vol. 319, The New England Journal of Medicine. 1988. p. 1701–6.
- 9. Leipzig RM, Cumming RG, Tinetti ME. Drugs and falls in older people: a systematic review and meta-analysis: II. Cardiac and analgesic drugs. J Am Geriatr Soc. 1999;47:40–50.
- 10. Leipzig RM, Cumming RG, Tinetti ME. Drugs and falls in older people: a systematic review and meta-analysis: I. Psychotropic drugs. J Am Geriatr Soc. 1999;47:40–50.
- 11. Cumming RG. Epidemiology of medication-related falls and fractures in the elderly. Drugs Aging. 1998 Jan;12(1):43–53.
- 12. Hartikainen S, Lönnroos E, Louhivuori K. Medication as a risk factor for falls: critical systematic review. J Gerontol A Biol Sci Med Sci. 2007 Oct;62(10):1172–81.
- 13. Woolcott JC, Richardson KJ, Wiens MO, Patel B, Marin J, Khan KM, et al. Meta-analysis of the impact of 9 medication classes on falls in elderly persons. Arch Intern Med. 2009 Nov;169(21):1952–60.
- 14. Seppala LJ, Petrovic M, Ryg J, Bahat G, Topinkova E, Szczerbińska K, et al. STOPPFall (Screening Tool of Older Persons Prescriptions in older adults with high fall risk): a Delphi study by the EuGMS Task and Finish Group on Fall-Risk-Increasing Drugs. Age Ageing. 2021;50(4):1189–99.
- 15. Seppala LJ, van de Glind EMM, Daams JG, Ploegmakers KJ, de Vries M, Wermelink AMAT, et al. Fall-Risk-Increasing Drugs: A Systematic Review and Meta-analysis: III. Others. J Am Med Dir Assoc. 2018 Apr;19(4):372.e1-372.e8.
- 16. Seppala LJ, Wermelink AMAT, de Vries M, Ploegmakers KJ, van de Glind EMM, Daams JG, et al. Fall-Risk-Increasing Drugs: A Systematic Review and Meta-Analysis: II.

- Psychotropics. J Am Med Dir Assoc. 2018 Apr;19(4):371.e11-371.e17.
- 17. de Vries M, Seppala LJ, Daams JG, van de Glind EMM, Masud T, van der Velde N. Fall-Risk-Increasing Drugs: A Systematic Review and Meta-Analysis: I. Cardiovascular Drugs. J Am Med Dir Assoc. 2018 Apr;19(4):371.e1-371.e9.
- 18. Seppala LJ, van der Velde N, Masud T, Blain H, Petrovic M, van der Cammen TJ, et al. EuGMS Task and Finish group on Fall-Risk-Increasing Drugs (FRIDs): Position on Knowledge Dissemination, Management, and Future Research. Drugs Aging. 2019 Apr;36(4):299–307.
- 19. Gade GV, Jørgensen MG, Ryg J, Masud T, Jakobsen LH, Andersen S. Development of a multivariable prognostic PREdiction model for 1-year risk of FALLing in a cohort of community-dwelling older adults aged 75 years and above (PREFALL). BMC Geriatr. 2021 Jun;21(1):402.
- 20. Gade GV, Jørgensen MG, Ryg J, Masud T, Andersen S. Development of a Multivariable Prognostic PREdiction Model for 1-year Risk of FALLing in Community-dwelling Older Adults in a Non-clinical Setting (PROTOCOL) [Internet]. [cited 2021 Oct 5]. Available from: https://clinicaltrials.gov/ct2/show/NCT03608709
- 21. von Elm E, Altman DG, Egger M, Pocock SJ, Gøtzsche PC, Vandenbroucke JP. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. Lancet [Internet]. 2007 Oct 20;370(9596):1453–7. Available from: https://doi.org/10.1016/S0140-6736(07)61602-X
- 22. Sundhedsstyrelsen. Forebyggelse på ældreområdet håndbog til kommunerne [Internet]. 2015 [cited 2021 Oct 5]. Available from: https://www.sst.dk/-/media/Udgivelser/2015/Forebyggelse-på-ældreområdet---håndbog-til-kommunerne/Forebyggelse-på-ældreområdet,-d-,-Håndbog-til-kommunerne.ashx?la=da&hash=74B7EC7B72EA05AD8BE434F866BFA586AC36BF9B
- 23. Sørensen G V., Jørgensen MG, Ryg J, Masud T, Andersen S. Development, feasibility, acceptability, and adjustment of a portable, multifactorial falls risk test battery for community-dwelling older adults. Cogent Med [Internet]. 2019;6(1):1674099. Available from: https://doi.org/10.1080/2331205X.2019.1674099
- 24. Munck LK, Hansen KR, Grethe Mølbak A, Balle H, Kongsgren S. The use of shared medication record as part of medication reconciliation at hospital admission is feasible. Dan Med J. 2014;61(5):1–5.
- 25. Jehu DA, Davis JC, Falck RS, Bennett KJ, Tai D, Souza MF, et al. Risk factors for recurrent falls in older adults: A systematic review with meta-analysis. Maturitas [Internet]. 2021 Feb;144(November 2020):23–8. Available from: https://doi.org/10.1016/j.maturitas.2020.10.021
- 26. Lord SR, Menz HB, Sherrington C. Falls in Older People. In: Osteoporosis in Clinical Practice: A Practical Guide for Diagnosis and Treatment [Internet]. London: Springer London; 2004. p. 93–9. Available from: https://doi.org/10.1007/978-0-85729-402-9\_12
- 27. Pluijm SMF, Smit JH, Tromp EAM, Stel VS, Deeg DJH, Bouter LM, et al. A risk profile for identifying community-dwelling elderly with a high risk of recurrent falling: Results of a 3-year prospective study. Osteoporos Int. 2006;17(3):417–25.

- 28. Delbaere K, Close JCT, Heim J, Sachdev PS, Brodaty H, Slavin MJ, et al. A multifactorial approach to understanding fall risk in older people. J Am Geriatr Soc. 2010;58(9):1679–85.
- 29. Rossat A, Fantino B, Nitenberg C, Annweiler C, Poujol L, Herrmann FR, et al. Risk factors for falling in community-dwelling older adults: which of them are associated with the recurrence of falls? J Nutr Health Aging. 2010 Nov;14(9):787–91.
- 30. Kempen GIJM, Yardley L, Van Haastregt JCM, Zijlstra GAR, Beyer N, Hauer K, et al. The Short FES-I: A shortened version of the falls efficacy scale-international to assess fear of falling. Age Ageing. 2008;37(1):45–50.
- 31. Quach L, Galica AM, Jones RN, Procter-Gray E, Manor B, Hannan MT, et al. The nonlinear relationship between gait speed and falls: the Maintenance of Balance, Independent Living, Intellect, and Zest in the Elderly of Boston Study. J Am Geriatr Soc. 2011 Jun;59(6):1069–73.
- 32. Stenhagen M, Nordell E, Elmståhl S. Falls in elderly people: a multifactorial analysis of risk markers using data from the Swedish general population study "Good ageing in Skåne". Aging Clin Exp Res. 2013 Apr;25(1):59–67.
- 33. Stenhagen M, Ekström H, Nordell E, Elmståhl S. Falls in the general elderly population: a 3-and 6- year prospective study of risk factors using data from the longitudinal population study "Good ageing in Skane". BMC Geriatr. 2013 Aug;13:81.
- 34. Dellasega CA, Lacko L, Singer H, Salerno F. Telephone screening of older adults using the Orientation-Memory-Concentration test. Geriatr Nurs. 2001;22(5):253–7.
- 35. Andreasen J, Sørensen EE, Gobbens RJJ, Lund H, Aadahl M. Danish version of the Tilburg Frailty Indicator--translation, cross-cultural adaption and validity pretest by cognitive interviewing. Arch Gerontol Geriatr. 2014;59(1):32–8.
- 36. Saliba D, Elliott M, Rubenstein LZ, Solomon DH, Young RT, Kamberg CJ, et al. The Vulnerable Elders Survey: a tool for identifying vulnerable older people in the community. J Am Geriatr Soc. 2001 Dec;49(12):1691–9.
- 37. Treves N, Perlman A, Kolenberg Geron L, Asaly A, Matok I. Z-drugs and risk for falls and fractures in older adults-a systematic review and meta-analysis. Age Ageing. 2018 Mar;47(2):201–8.
- 38. Yoshikawa A, Ramirez G, Smith ML, Foster M, Nabil AK, Jani SN, et al. Opioid Use and the Risk of Falls, Fall Injuries and Fractures among Older Adults: A Systematic Review and Meta-Analysis. J Gerontol A Biol Sci Med Sci. 2020 Sep;75(10):1989–95.
- 39. Lamb SE, Jørstad-Stein EC, Hauer K, Becker C. Development of a common outcome data set for fall injury prevention trials: The Prevention of Falls Network Europe consensus. J Am Geriatr Soc. 2005;53(9):1618–22.